CLINICAL TRIAL: NCT06477120
Title: A Pilot Study of Time-restricted Eating Among Pregnant Females With Severe Obesity
Brief Title: Time-restricted Eating Among Pregnant Females With Severe Obesity
Acronym: TRE-Preg
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lisa Tussing-Humphreys, Professor, Kinesiology and Nutrition, PhD, MS, RD, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-0138; 5R01DK136085-02 (NIH)
Record Dates: First submitted 2024-05-30; First posted 2024-06-27 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Obesity, Morbid; Time Restricted Eating; Pregnancy Weight Gain
MeSH Terms: conditions — Obesity, Morbid; Intermittent Fasting; Gestational Weight Gain

STUDY DESIGN:
Intervention Model Description: 1:1 allocation ratio. Randomization will be stratified by participant age (18-30 and 31-44 years old).
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-restricted eating (Experimental): Participants randomized to the time-restricted eating arm will be instructed to eat ad libitum during an 8-hr window daily 11am - 7pm in the 2nd trimester and 10-hr eating window from 10am - 8pm in the 3rd trimester and abstain from caloric foods and beverages for the remaining 14-16 hours. During the eating window there will be no restrictions on types or quantities of foods consumed. Moreover, participants will not be required to monitor calorie intake during the ad libitum eating period. During the fasting period, participants will be encouraged to drink plenty of water and will be allowed to consume calorie-free beverages.
  Interventions: Behavioral: Time Restricted Eating
- Enhanced Standard Care (No Intervention): The standard care arm will not receive diet-related counseling. Participants will meet with study staff weekly to record health changes and to transmit weight through the text messaging platform. The remote videoconferencing visits will occur at the same day and time each week. Standard care participants will attend the in-person research data collection visits. Participants will be asked to maintain current (baseline) level of physical activity throughout the intervention.

INTERVENTIONS:
Behavioral: Time Restricted Eating — The time-restricted eating arm will be instructed to eat ad libitum during an 8-hr window daily (10am - 6pm OR 11am - 7pm) in the 2nd trimester and 10-hr eating window from (9am - 7pm OR 10am - 8pm) in the 3rd trimester and abstain from caloric foods and beverages for the remaining 14-16 hours.
  Arms: Time-restricted eating

SUMMARY:
In the United States, a body mass index (BMI) of at least 35.0 kg/m2 affects about 15% of women of reproductive age. Severe obesity is a significant predictor of adverse perinatal outcomes including gestational diabetes mellitus, pre-eclampsia, premature birth, and at its most severe, fetal death, birth defects and a three-fold greater risk of maternal mortality. Observational studies suggest weight maintenance and even modest body fat loss and altering the maternal metabolic milieu (availability of glucose and lipids) in the gestational period may be important to reducing perinatal health risks among pregnant females with severe obesity. The proposed research aims to assess time-restricted eating in the 2nd and 3rd trimesters of pregnancy to explore the effects on maternal weight, and perinatal health outcomes compared to standard clinical care.

DETAILED DESCRIPTION:
Severe obesity is a contributor to adverse perinatal outcomes. The prevalence of severe obesity is on the rise in the United States (U.S.), having increased from 6.4% of the adult population in 2011-2012 to just over 9% of adults in 2017-2018. The prevalence of severe obesity among reproductive age females is approximately 10%. This is an alarming statistic given severe obesity is a predictor of adverse perinatal outcomes including gestational diabetes mellitus, preeclampsia, premature birth (both spontaneous and medically indicated), and at its most severe, fetal death, birth defects, and a three-fold greater risk of maternal mortality. Observational studies suggest weight maintenance and even modest body fat loss and altering the maternal metabolic milieu (availability of glucose and lipids) in the gestational period may be important to reducing perinatal health risks among pregnant females with severe obesity. Existing lifestyle interventions (calorie control/dietary pattern changes/physical activity) have showed modest effects on attenuating excess gestational weight gain and modest effects on perinatal health outcomes among pregnant females with obesity. Time- restricted eating, where an individual simply watches the clock and consumes calories within a particular eating window, is a simple and highly accessible eating pattern that has the potential to minimize gestational weight gain, reduce excess glucose and lipids, and improve metabolic health among pregnant females with severe obesity all of which could translate to improved perinatal health outcomes. Yet there are no clinical trials of time-restricted eating in pregnancy. The investigators aim to test the safety, feasibility, and acceptability of time-restricted eating among 60 pregnant females with severe obesity. The investigators will examine time-restricted eating safety, feasibility and acceptability (8-hr eating window in the 2nd trimester & 10-hr eating window in the 3rd trimester), and explore its effects on weight, cardiometabolic risk markers and perinatal health outcomes vs. Standard Care. The intervention will begin between 14 - < = 20 weeks gestational age and continue through admission for labor and delivery. The study will involve weekly meetings with a nutritionist, and research visits at baseline (~17 weeks gestational age), 27-29 weeks gestational age and 35-37 weeks gestational age as well as monthly check-ins for maternal and fetal health monitoring. Maternal and neonatal data from labor and delivery will also be collected from electronic health records. Glucose will be continuously monitored for 10 days at 20 weeks gestational age and 34 weeks gestational age (optional). The goal of our work is to reduce and prevent adverse perinatal outcomes among pregnant females with severe obesity. Given the relative simplicity of time-restricted eating it can be easily disseminated in clinic demonstrating its strong potential for wide-scale public health impact.

ELIGIBILITY:
Inclusion criteria:

* Female based on sex assigned at birth
* Preconception body mass index (BMI) 35.0 - 60 kg/m2
* Singleton pregnancy
* Age 18-44 years old
* 14 - < = 20 weeks gestational age
* Fluency in English to provide consent and complete study procedures
* Ability to provide informed consent
* Cleared by study doctor and the obstetrician/mid-wife provider to participate
* Access to a smartphone to complete intervention procedures

Exclusion criteria:

* Deemed medically high risk
* Multiple pregnancy (e.g., twins)
* Type 1 or 2 diabetes mellitus
* Early gestational diabetes (diagnosed at < = to17 weeks gestational age through an oral glucose tolerance test)
* Currently eating ≤ 12 hours daily
* Autoimmune disorder (e.g., rheumatoid arthritis)
* iron deficiency anemia
* Inflammatory bowel disease
* Previous spontaneous preterm birth
* History of bariatric surgery
* Night shift work
* Currently incarcerated
* Eating disorder

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-11-29 (Estimated)

PRIMARY OUTCOMES:
Recruitment Feasibility | From 6 months through 32 months (the funding period is 36 months)
  ≥ 30% of those approached enroll
Trial safety - Maternal Complete Blood Count | Baseline (14-20 weeks gestational age) and monthly through labor and delivery, about 6 months
  % and n with abnormal results by study arm
Trial safety - Non-stress Test for Fetal Safety | 29-31 weeks gestational age and 35-37 weeks gestational age
  Measured with a fetal monitor to examine baby's heart rate over time (usually 20 to 30 minutes, but sometimes up to an hour) % and n with abnormal results by study arm
Intervention acceptability | 25-27 weeks gestational age and 35-37 weeks gestational age
  Semi-structured interviews
Research visit feasibility | Baseline, 25-27 weeks gestational age and 35-37 weeks gestational age
  Number of data collection visits completed with >=80% completed at each timepoint and completeness of data
Intervention (TRE) session feasibility | Weekly from baseline through labor and delivery, about 6 months
  Number and % of intervention sessions completed by TRE participants
TRE adherence | Daily from enrollment to labor and delivery (TRE arm only), about 6 months
  Response rate to daily text message regarding eating start and stop time to determine adherence to the eating window goal is >= 80% adherence on days reported
Trial safety - Maternal health checks | Weekly from baseline to labor and delivery, about 6 months, % and n for health events reported by study arm
  Weekly maternal health checks via videoconference in TRE and control group that is verified with electronic health record
Trial safety - Maternal outcomes | Labor and delivery
  Data obtained from the participant's electronic health record (gestational age at delivery, gestational diabetes, gestational hypertension, preeclampsia, c-section, spontaneous pre-term birth, iron deficiency anemia) % and n with abnormal results by study arm
Trial safety - Neonatal outcomes | Labor and delivery
  Data obtained from the participant's electronic health record (small or large for gestational age, neonatal intensive care admission, jaundice, APGAR score) % and n with abnormal results by study arm
Trial Retention | 35-37 week gestational age
  n and % of women retained through the final in-person data collection with >= 80% retained

SECONDARY OUTCOMES:
Maternal Body Weight | Baseline (14-20 weeks), 25-27 weeks gestational age, 35-37 weeks gestational age
  Body weight in kilograms
Maternal Fasting Blood Glucose | Baseline (14-20 weeks gestational age), 25-27 weeks gestational age, 35-37 weeks gestational age
  Measured in serum
Maternal Fasting Insulin | Baseline (14-20 weeks gestational age), 25-27 weeks gestational age, 35-37 weeks gestational age
  Measured in serum
Maternal Fasting Blood Lipids | Baseline (14-20 weeks gestational age), 25-27 weeks gestational age, 35-37 weeks gestational age
  Cholesterol and triglycerides
Maternal C-reactive protein | Baseline (14-20 weeks gestational age), 25-27 weeks gestational age, 35-37 weeks gestational age
  Measured in plasma
Maternal Systolic Blood Pressure | Baseline (14-20 weeks gestational age), 25-27 weeks gestational age, 35-37 weeks gestational age
  Measured with participant in a seated position using an automated cuff
Maternal Diastolic Blood Pressure | Baseline (14-20 weeks), 25-27 weeks gestational age, 35-37 weeks gestational age
  Measured with participant in a seated position using an automated cuff
Maternal Hb A1c | Baseline (14-20 weeks gestational age), 25-27 weeks gestational age, 35-37 weeks gestational age
  Measured from whole blood

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago College of Applied Health Sciences, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No